CLINICAL TRIAL: NCT06745934
Title: Healthy Minds for Pre-Service Teachers
Brief Title: Strengthening Health and Insight in New Educators
Acronym: SHINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Summer Braun, Assistant Professor, University of Alabama, Tuscaloosa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-01-7242; R15MH134225 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Anxiety Symptoms; Depressive Symptoms
Keywords: Healthy Minds Program; mindfulness-based intervention; app; pre-service teachers; mental health
MeSH Terms: conditions — Anxiety Disorders; Depression; Alzheimer Disease; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Business as Usual (No Intervention): Participants in this arm will continue with daily life as usual.
- Healthy Minds Program (Experimental): Participants in this arm engage with the Healthy Minds Program app.
  Interventions: Behavioral: Healthy Minds Program

INTERVENTIONS:
Behavioral: Healthy Minds Program — Participants in this arm engage with the Healthy Minds Program app/
  Arms: Healthy Minds Program

SUMMARY:
Teachers are at notable risk for depression and anxiety. The present study tests an app-based mindfulness intervention for teachers in their final year of training with the goal of preventing the deterioration of their mental health during the transition into the classroom. The project will strengthen the research environment at the University of Alabama and will involve undergraduate research assistants in each step of the research process.

DETAILED DESCRIPTION:
Mental health concerns in teachers have escalated since the onset of the pandemic, and the deterioration of mental health can begin as early as the teacher training period. Accessible and scalable programs that prepare teachers for the stress of the profession are urgently needed to prevent the deterioration of mental health and its attendant consequences. The goal of this longitudinal project is to test the feasibility and acceptability, utility, and candidate mechanisms of an accessible, mobile health, mindfulness-based intervention, the Healthy Minds Program (HMP), to equip teachers in training ("pre-service teachers"; i.e., university students majoring in education) with skills necessary to maintain their mental health as they transition into the classroom. The project addresses three specific aims. Aim 1: a) Assess the feasibility and acceptability of the HMP for pre-service teachers and b) identify barriers and facilitators to program acceptability. Aim 2: Determine the utility of the HMP for preventing depression and anxiety (main outcomes) and turnover intentions (secondary outcome). Aim 3: Examine HMP effects on candidate mechanisms, and the effect of mechanisms on outcomes. The results of this project will provide critical insight into the potential for the HMP to scale up for widespread use in pre-service teacher training programs. Importantly, the project will provide a unique opportunity for undergraduate research at the University of Alabama, and will strengthen the research environment by involving undergraduate research assistants in each step of the research process.

ELIGIBILITY:
Inclusion Criteria:

* Students in Block 3 will be invited to participate in the study.

Exclusion Criteria:

* Students who are not in Block 3 will be excluded. Participants experiencing suicidal ideations at baseline and deemed via the clinical risk assessment procedure to be at moderate or high risk of suicide will be excluded from the study after baseline, and prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression - Short Form 8b | Participants will report on depression at baseline, post-intervention (3 months after baseline), 3-month follow-up , and 12-month follow-up.
  Participants will self-report on depression. Each of the 8 items is rated on 1 (1 = Never) to 5 (5 = Always) scale. Responses will be summed to create the raw scale score. Higher values indicate greater symptoms of depression (i.e., a worse outcome).
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety - Short Form 7a | Participants will report on anxiety at baseline, post-intervention (3 months after baseline), 3-month follow-up, and 12-month follow-up.
  Participants will self-report on anxiety. Each of the 7 items is rated on 1 (1 = Never) to 5 (5 = Always) scale. Responses will be summed to create the raw scale score. Higher values indicate greater symptoms of anxiety (i.e., a worse outcome).

SECONDARY OUTCOMES:
Turnover Intentions | Participants will report turnover intentions at 3-month follow-up, and 12-month follow-up.
  Participants will self-report on their intentions to leave their job.

OTHER OUTCOMES:
Teaching Quality: edTPA | edTPA scores will be collected immediately after the intervention.
  Performance-based assessment of teaching quality required for teacher certification. Higher scores indicate greater teaching quality.
Teaching Quality: Candidate Preservice Assessment of Student Teaching (CPAST) | CPAST scores will be collected immediately after the intervention.
  Summative assessment of pre-service teachers' teaching quality during the semester-long student teaching experience. Higher scores indicate greater teaching quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama, Tuscaloosa, Alabama, United States